CLINICAL TRIAL: NCT04921644
Title: Longitudinal Investigation of Cancer-related Fatigue and Its Treatment (LIFT Project)
Status: Active, not recruiting | Type: Observational
Sponsor: German Cancer Research Center (Other)
Collaborators: Wuerzburg University Hospital (Other); Baden-Württemberg Cancer Registry (Unknown); German Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: LIFT project
Record Dates: First submitted 2021-04-09; First posted 2021-06-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Cancer-related Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patient cohort: Newly diagnosed patients with colon, rectum, liver, pancreas or lung cancer, malignant melanoma, breast or other gynecological cancers, prostate, kidney, bladder or thyroid gland cancer, non-Hodgkin lymphoma or leukemia recruited approximately 6 months after diagnosis and followed up to 2 years post-diagnosis. No intervention.

SUMMARY:
The LIFT project aims to thoroughly investigate the current status of health care in Germany regarding cancer-related fatigue from the institutional, professionals' and patients' perspective.

DETAILED DESCRIPTION:
The LIFT project aims to thoroughly investigate the current status of health care in Germany regarding fatigue from the institutional, professionals', and patients' perspective. With a multimodal approach including a comprehensive assessment of fatigue management and support offered by different institutions (uncertified hospitals, uncertified oncological practices, counselling units, certified cancer centers; n=350), a survey and qualitative interviews among practicing physicians ("Niedergelassene Ärzte"), hospital physicians, practicing psychotherapists with psycho-oncological focus, psycho-oncologists at hospitals, nurses at certified cancer centers and nurses at other hospitals (n=420), and a longitudinal clinical study among cancer patients (n=1400) as well as two focus groups with patient representatives (each n=6), the characteristics, patterns, and potential effects or shortcomings of the current fatigue management will be investigated. Furthermore, factors associated with patients' and health care professionals' knowledge about fatigue will be examined.

Concerning the longitudinal clinical study assessing the patients' perspective, online or paper-based questionnaires on socio-demographic, clinical and patient reported outcomes will be sent to the patients 6,9,12 and 24 months after diagnosis. Moreover, detailed data on screening, diagnosis and counseling as well as therapies offered and administered to reduce fatigue will be surveyed, as well as the patients' state of knowledge, perception and prevailing needs regarding fatigue. Tumor and cancer therapy data will be extracted from the Epidemiological Cancer Registry.

The results of the LIFT project shall provide a basis to identify and overcome shortcomings in the actual fatigue management in Germany, and, to eventually ameliorate this severe burden in cancer patients and survivors.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Newly diagnosed with a primary tumor of one of the following malignant neoplasms: colon (C18), rectum (C19-20), liver (C22), pancreas (C25), lung (C33-34), malignant melanoma (C43), breast (C50, only female), cervix (C53), endometrium (C54.1), ovaries (C56), prostate (C61), kidney (C64), bladder (C67), thyroid gland (C73), non-Hodgkin lymphoma (C82-88), leukemia (C91-C95)
* Having received or receiving at enrolment at least one of the following treatments: chemotherapy, radiotherapy, hormone therapy, targeted or immune therapy
* Able to understand and follow the study protocol

Exclusion Criteria:

* Carcinoma in situ
* Any additional malignant or unclear neoplasm before or since time of diagnosis of the considered primary tumor, except unspecified neoplasm of skin (C44)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with colon, rectum, liver, pancreas or lung cancer, malignant melanoma, breast or other gynecological cancers, prostate, kidney, bladder or thyroid gland cancer, non-Hodgkin lymphoma or leukemia.
Sampling Method: Probability Sample
Enrollment: 1183 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2023-01-07 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue severity | 6 months after diagnosis to 2 years post-diagnosis
  assessed by EORTC QLQ-FA12 (European Organisation for Research and Treatment of Cancer Quality of Life Fatigue Questionnaire). The items are rated on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much) with higher scores meaning a higher level of fatigue.
Impact of fatigue | 6 months after diagnosis to 2 years post-diagnosis
  assessed by the Brief Fatigue Inventory (BFI). The BFI consists of an 11-point numerical rating scale ranging from 0 (no fatigue) to 10 (as bad as you can imagine) with higher scores signifying higher intensity and impairment.
State of fatigue management | 6 months after diagnosis to 2 years post-diagnosis
  Questionnaire assessing the adherence to the National Comprehensive Cancer Network (NCCN) guidelines regarding management of cancer-related fatigue.
Knowledge, attitudes and beliefs regarding cancer-related fatigue | 6 months after diagnosis to 2 years post-diagnosis
  Questionnaire assessing knowledge, attitudes and beliefs regarding cancer-related fatigue. The knowledge score consists of fatigue-related statements that should be rated as either right, wrong, or "dont know". The attitudes scale is composed of statements that should be rated on a 4-point likert scale. Higher scores indicate a greater agreement to the particular statement.

SECONDARY OUTCOMES:
Quality of life functions and symptoms | 6 months after diagnosis to 2 years post-diagnosis
  assessed by EORTC QLQ-C30 and 5 additional items derived according to the EORTC scoring manual assessing symptoms of fever, hot flashes, night sweat, polyneuropathy and distress of dependents caused by the diagnosis are added. The items are rated on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much). A higher score corresponds to a higher level of symptoms/problems.
Sleep problems | 6 months after diagnosis to 2 years post-diagnosis
  assessed by Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of open and closed questions regarding characteristics of sleep and sleep quality. Some items are rated on a 4-point likert scale with higher scores meaning more sleep problems.
Depression | 6 months after diagnosis to 24 months post-diagnosis
  assessed by Patient Health Questionnaire (PHQ-9). The items are rated on a 4-point scale ranging from 0 (not at all) to 3 (most of the time). A sum score is calculated, with higher scores meaning a higher level of depressive symptoms.
Body mass index | 6 months, 12 months and 24 months post-diagnosis
  calculated from weight and height
Total physical activity | 6 months, 12 months and 24 months post-diagnosis
  assessed by a questionnaire regarding walking, cycling and exercise behavior
Return to work | 6 months, 12 months and 24 months post-diagnosis
  assessed by questions regarding occupational issues
Anxiety | assessed 6 months after diagnosis to 24 months after diagnosis
  assessed by the Generalized Anxiety Disorder Questionnaire (GAD-7). The items are rated on a 4-point scale ranging from 0 (not at all) to 3 (most of the time). A sum score (ranging from 0 to 21) is calculated, with higher scores meaning a higher level of symptomatology.
Supportive Care Needs | assessed at t2 9 months post-diagnosis
  assessed by the Supportive Care Needs Survey (SCNS-SF-34). The scale ranges from 1 (not applicable) to 5 (high need) with higher scores meaning a higher need of support.
Social Support | at t1 (6 months post-diagnosis) and t3 (12 months post-diagnosis)
  assessed by the Illness-specific Social Support Scale (ISSS, German Version) among cancer patients. The 8 items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (always). Sum scores for the items 1,3,6 and 8 (positive support) as well as for the items 2,4,5 and 7 (detrimental interaction) are calculated with higher scores meaning higher levels of positive support and detrimental interaction respectively.
Loneliness | at t1 (6 months post-diagnosis) and t4 (24 months post-diagnosis)
  assessed by three items of the University of California, Los Angeles (UCLA)-loneliness-scale. The response categories are 1 (hardly ever), 2 (some of the time) and 3(often). A sum score is calculated with higher scores meaning a higher level of loneliness.
Resilience | assessed at t1 6 months post-diagnosis
  assessed by the Brief Resilience Scale (BRS). The six items are rated on a 5-point Likert-scale ranging from 1 (strongly disagree) to 5 (strongly agree). After reversing the coding of inverted items 2,4 and 6, the mean of the six items is calculated with higher scores meaning a higher level of resilience.
Patient Activation | at t2 (9 months post-diagnosis)
  assessed by the Patient Activation Measure (PAM-13). Patients are supposed to rate their level of agreement to 13 statements on a 4-point-scale. A higher score corresponds to a higher level of patient activation.
Posttraumatic growth | at t4 (24 months post-diagnosis)
  assessed by Posttraumatic Growth Inventory (PTGI). The items are rated on a 6-point Likert scale ranging from 1 (not at all) to 6 (very strongly) with higher scores indicating a higher level of posttraumatic growth.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Steindorf, Prof. Dr., Principal Investigator — German Cancer Research Center, Division of Physical Activity, Prevention and Cancer; Martina E. Schmidt, Dr., Principal Investigator — German Cancer Research Center, Division of Physical Activity, Prevention and Cancer; Imad Maatouk, Prof. Dr., Principal Investigator — Psychosomatics, Psychotherapy and Psycho-Oncology, Medical Hospital II, University Hospital Wuerzburg
Locations (1):
- German Cancer Research Center, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wagner AS, Milzer M, Schmidt ME, Kiermeier S, Maatouk I, Steindorf K. Nurses' Knowledge of Cancer-Related Fatigue and the Coverage of This Subject in Nursing Training: A Cross-Sectional Study. J Nurs Res. 2025 Apr 1;33(2):e379. doi: 10.1097/jnr.0000000000000666. PMID 40162696
- [Derived] Wagner AS, Wehlen L, Milzer M, Schmidt ME, Kiermeier S, Maatouk I, Steindorf K. Physicians' perspectives on cancer-related fatigue management and their suggestions for improvements in medical training: a cross-sectional survey study in Germany. Support Care Cancer. 2024 Nov 14;32(12):788. doi: 10.1007/s00520-024-08978-2. PMID 39537876
- [Derived] Milzer M, Wagner AS, Schmidt ME, Maatouk I, Hermann S; Cancer Registry of Baden-Wurttemberg; Kiermeier S, Steindorf K. Patient-physician communication about cancer-related fatigue: a survey of patient-perceived barriers. J Cancer Res Clin Oncol. 2024 Jan 25;150(2):29. doi: 10.1007/s00432-023-05555-8. PMID 38270814
- [Derived] Milzer M, Wagner AS, Steindorf K, Kiermeier S, Schmidt ME, Maatouk I. Psycho-oncologists' knowledge of cancer-related fatigue and the targets for improving education and training: results from a cross-sectional survey study. Support Care Cancer. 2023 Jun 23;31(7):412. doi: 10.1007/s00520-023-07882-5. PMID 37351639